CLINICAL TRIAL: NCT02564120
Title: North Carolina Prostate Cancer Comparative Effectiveness & Survivorship Study (NC ProCESS)
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: UNC-10-1483
Record Dates: First submitted 2015-08-26; First posted 2015-09-30 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Cancer of Prostate; Cancer of the Prostate; Prostate Cancer; Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
NC ProCESS is a cohort of patients from diverse backgrounds diagnosed with early prostate cancer, who were enrolled from January 2011-June 2013. These patients were recruited throughout North Carolina, and also in partnership with institutions across the country. Patients enrolled before they start treatment, and are then followed prospectively through treatment and then afterwards. This observational study collects information on quality of life, cancer control, and health care received inclusive of treatment and management of subsequent effects including complications and recurrence. The objective of this study is to examine comparative outcomes among different modern prostate cancer treatment options in this cohort of patients.

DETAILED DESCRIPTION:
Localized prostate cancer treatment options is consistently a "highest priority" comparative effectiveness research (CER) topic according to the Institute of Medicine, Agency for Healthcare Research and Quality (AHRQ), and other summary reports. Patients urgently need information on the comparative outcomes of modern treatment options to guide decision-making for this disease that causes significant burden based on its high prevalence, mortality and treatment effects on quality of life. The status quo as it pertains to prostate cancer is significant overtreatment causing potential patient harm, rapid diffusion of new/expensive technologies without proven benefit and patients lacking high quality research evidence to balance direct-to-consumer advertising and guide individualized decision-making.

NC ProCESS is a population-based cohort designed specifically to address well-described knowledge gaps. It was designed in close collaboration with the unique AHRQ consortium stakeholder group, which included representatives from patients, clinicians and policymakers. Stakeholders helped define study design to emphasize "real-world" patients and select patient-centered and relevant outcomes, and have been involved throughout assembly of this patient cohort. The diverse cohort is well-represented by "hard to reach" patients; enrollment before treatment avoids biases with participation and recall. As clinical trials are not feasible to address the central questions in prostate cancer CER, this prospective study will yield the highest level of evidence to inform patients and other stakeholders. With an assembled cohort, this study is necessary to examine comparative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed, histologically-proven, localized prostate adenocarcinoma.
* Completion of baseline interview prior to initiating therapy.
* Patient ability to complete study interview: no cognitive impairment, language or hearing problems.
* Not diagnosed with prostate cancer through transurethral resection of the prostate (TURP).
* Age 35-80.
* English speaking.
* Has telephone.

Exclusion Criteria:

* Initiation of treatment for prostate cancer prior to completion of baseline interview.
* Cognitive impairment.
* Hearing problems.
* Inability to speak or understand English.

Ages: 35 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly-diagnosed, early stage (localized, non-metastatic) prostate cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 1556 (Actual)
Dates: Start 2011-01; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NC ProCESS Cohort: NC ProCESS is a cohort of patients with early prostate cancer, who were enrolled from January 2011-June 2013. These patients were recruited throughout North Carolina, and also in partnership with institutions across the country. Patients enrolled before they started treatment, and were then followed prospectively.
Period: Overall Study
Arm/Group | NC ProCESS Cohort
Started | 1556
Completed | 1110
Not Completed | 446
Not completed — Did not return release forms | 160
Not completed — Death | 58
Not completed — Withdrawal by Subject | 204
Not completed — Other medical condition | 24

BASELINE CHARACTERISTICS:
Population: The analytic cohort comprised 1413 men who completed baseline survey information and either underwent active surveillance (n=390, 27.6%) or received treatment with SBRT (n=104, 7.4%), radical prostatectomy (n=547, 38.7%), conventional fractionation external beam radiation therapy (EBRT; n=247, 17.5%), or brachytherapy (n=125, 8.8%).
Groups:
- Active Surveillance: Men placed on active surveillance (i.e., did not receive immediate treatment)
- SBRT: Men who received stereotactic body radiation therapy
- Radical Prostatectomy: Men treated with radical prostatectomy (i.e., surgery)
- EBRT: Men treated with external beam radiation therapy
- Brachytherapy: Men treated with brachytherapy
- Total: Total of all reporting groups
Arm/Group | Active Surveillance | SBRT | Radical Prostatectomy | EBRT | Brachytherapy | Total
Number analyzed (Participants) | 390 | 104 | 547 | 247 | 125 | 1413
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.5) | 65.3 (6.8) | 61.1 (7.0) | 66.8 (7.1) | 64.6 (7.3) | 64.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 390 | 104 | 547 | 247 | 125 | 1413
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 287 | 97 | 382 | 153 | 90 | 1009
  African American | 97 | 3 | 143 | 83 | 33 | 359
  Other | 6 | 4 | 22 | 11 | 2 | 45
Region of Enrollment [Number; unit: participants]
  United States | 390 | 104 | 547 | 247 | 125 | 1413

OUTCOME MEASURES:

1. Primary Outcome: Cancer-specific Quality of Life
Description: Prostate Cancer Symptom Indices (PCSI) - measures treatment-related morbidity and adverse effects and is comprised of 4 functional scales measuring Sexual Dysfunction, Bowel Problems, Urinary Incontinence, and Urinary Obstruction/Irritation. Four parallel distress indices measure distress from symptoms. In each index, patient answers are converted to a score from 0 (no symptom/distress) to 100 (maximum symptoms/distress). A 5-10 point difference in QOL is considered "clinically meaningful."
Time Frame: 4 years
Population: We analyzed data from NC ProCESS, a population-based, prospective prostate cancer patient cohort. The analytic cohort were men who completed baseline survey info & either underwent active surveillance or received initial treatment with stereotactic body radiation therapy, radical prostatectomy, external beam radiation therapy, or brachytherapy.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Active Surveillance: Patients placed on active surveillance following diagnosis of prostate cancer. Active surveillance was defined with medical records stating this as the plan.
- Stereotactic Body Radiation Therapy: Patients who received initial treatment with stereotactic body radiation therapy (SBRT).
- Radical Prostatectomy: Patients who received initial treatment with radical prostatectomy.
- External Body Radiation Therapy: Patients who received initial treatment with external body radiation therapy (EBRT).
- Brachytherapy: Patients who received initial treatment with brachytherapy.
Arm/Group | Active Surveillance | Stereotactic Body Radiation Therapy | Radical Prostatectomy | External Body Radiation Therapy | Brachytherapy
Number analyzed (Participants) | 390 | 104 | 547 | 247 | 125
score on a scale
  Sexual Dysfunction - Baseline | 44.7 [40.9 to 48.5] | 42.0 [34.7 to 49.3] | 35.9 [32.8 to 39.0] | 52.1 [47.2 to 57.0] | 44.9 [38.0 to 51.8]
  Sexual Dysfunction - 3-months: number analyzed (Participants) | 306 | 99 | 445 | 224 | 108
  Sexual Dysfunction - 3-months | 44.4 [40.0 to 48.8] | 42.1 [34.7 to 49.5] | 78.0 [75.5 to 80.5] | 65.2 [60.3 to 70.1] | 59.0 [52.3 to 65.7]
  Sexual Dysfunction - 12-months: number analyzed (Participants) | 282 | 96 | 419 | 206 | 97
  Sexual Dysfunction - 12-months | 48.2 [43.8 to 52.6] | 48.2 [40.7 to 55.7] | 70.8 [67.9 to 73.7] | 62.8 [57.8 to 67.8] | 59.3 [52.3 to 66.3]
  Sexual Dysfunction - 24-months: number analyzed (Participants) | 237 | 80 | 381 | 181 | 82
  Sexual Dysfunction - 24-months | 55.2 [50.4 to 60.0] | 48.8 [40.8 to 56.8] | 68.2 [65.0 to 71.4] | 64.9 [59.7 to 70.1] | 62.3 [54.7 to 69.9]
  Sexual Dysfunction - 36-months: number analyzed (Participants) | 209 | 75 | 330 | 145 | 67
  Sexual Dysfunction - 36-months | 50.9 [45.8 to 56.0] | 52.3 [43.7 to 60.9] | 68.6 [65.1 to 72.1] | 64.2 [58.5 to 69.9] | 63.7 [55.9 to 71.5]
  Sexual Dysfunction - 48-months: number analyzed (Participants) | 190 | 54 | 302 | 141 | 69
  Sexual Dysfunction - 48-months | 56.5 [51.1 to 61.9] | 53.9 [44.0 to 63.8] | 69.7 [66.0 to 73.4] | 66.1 [60.4 to 71.8] | 64.0 [55.7 to 72.3]
  Urinary Obstruction & Irritation - Baseline | 23.4 [22.0 to 24.8] | 22.9 [20.4 to 25.4] | 23.3 [22.1 to 24.5] | 24.2 [22.2 to 26.2] | 17.5 [15.7 to 19.3]
  Urinary Obstruction & Irritation - 3-months: number analyzed (Participants) | 306 | 99 | 445 | 224 | 108
  Urinary Obstruction & Irritation - 3-months | 23.2 [21.7 to 24.7] | 24.3 [21.7 to 26.9] | 27.0 [25.5 to 28.5] | 35.6 [33.0 to 38.2] | 40.3 [36.3 to 44.3]
  Urinary Obstruction & Irritation - 12-months: number analyzed (Participants) | 282 | 96 | 419 | 206 | 97
  Urinary Obstruction & Irritation - 12-months | 25.9 [24.1 to 27.7] | 29.5 [26.2 to 32.8] | 21.4 [20.1 to 22.7] | 25.3 [23.2 to 27.4] | 27.6 [24.3 to 30.9]
  Urinary Obstruction & Irritation - 24-months: number analyzed (Participants) | 237 | 80 | 381 | 181 | 82
  Urinary Obstruction & Irritation - 24-months | 25.1 [23.3 to 26.9] | 26.4 [23.3 to 29.5] | 19.4 [18.1 to 20.7] | 23.7 [21.6 to 25.8] | 26.9 [23.5 to 30.3]
  Urinary Obstruction & Irritation - 36-months: number analyzed (Participants) | 209 | 75 | 330 | 145 | 67
  Urinary Obstruction & Irritation - 36-months | 23.7 [21.9 to 25.5] | 22.8 [19.6 to 26.0] | 19.5 [18.2 to 20.8] | 22.5 [20.3 to 24.7] | 19.5 [16.7 to 22.3]
  Urinary Obstruction & Irritation - 48-months: number analyzed (Participants) | 190 | 54 | 302 | 141 | 69
  Urinary Obstruction & Irritation - 48-months | 24.3 [22.3 to 26.3] | 22.9 [19.9 to 25.9] | 19.2 [17.9 to 20.5] | 23.8 [21.5 to 26.1] | 22.2 [19.0 to 25.4]
  Urinary Incontinence - Baseline | 11.0 [8.9 to 13.1] | 8.3 [5.2 to 11.4] | 8.6 [7.1 to 10.1] | 14.1 [11.2 to 17.0] | 6.0 [3.4 to 8.6]
  Urinary Incontinence - 3-months: number analyzed (Participants) | 306 | 99 | 445 | 224 | 108
  Urinary Incontinence - 3-months | 12.3 [9.9 to 14.7] | 12.7 [9.1 to 16.3] | 44.0 [41.3 to 46.7] | 17.6 [14.2 to 21.0] | 15.1 [11.0 to 19.2]
  Urinary Incontinence - 12-months: number analyzed (Participants) | 282 | 96 | 419 | 206 | 97
  Urinary Incontinence - 12-months | 14.0 [11.4 to 16.6] | 15.2 [10.9 to 19.5] | 31.5 [29.0 to 34.0] | 18.7 [15.0 to 22.4] | 13.9 [9.9 to 17.9]
  Urinary Incontinence -24-months: number analyzed (Participants) | 237 | 80 | 381 | 181 | 82
  Urinary Incontinence -24-months | 18.6 [15.4 to 21.8] | 14.8 [10.0 to 19.6] | 29.7 [27.1 to 32.3] | 20.1 [16.3 to 23.9] | 16.3 [11.4 to 21.2]
  Urinary Incontinence - 36-months: number analyzed (Participants) | 209 | 75 | 330 | 145 | 67
  Urinary Incontinence - 36-months | 15.9 [12.8 to 19.0] | 15.1 [10.5 to 19.7] | 28.8 [26.0 to 31.6] | 20.4 [16.2 to 24.6] | 21.6 [15.7 to 27.5]
  Urinary Incontinence - 48-months: number analyzed (Participants) | 190 | 54 | 302 | 141 | 69
  Urinary Incontinence - 48-months | 19.9 [16.5 to 23.3] | 11.5 [6.8 to 16.2] | 30.8 [28.0 to 33.6] | 19.9 [15.6 to 24.2] | 16.5 [11.4 to 21.6]
  Bowel Problems - Baseline | 6.1 [5.3 to 6.9] | 5.5 [4.2 to 6.8] | 5.8 [5.1 to 6.5] | 7.5 [6.2 to 8.8] | 4.8 [3.5 to 6.1]
  Bowel Problems - 3-months: number analyzed (Participants) | 306 | 99 | 445 | 224 | 108
  Bowel Problems - 3-months | 7.1 [6.0 to 8.2] | 5.6 [4.3 to 6.9] | 7.1 [6.3 to 7.9] | 12.6 [10.5 to 14.7] | 9.0 [7.1 to 10.9]
  Bowel Problems - 12-months: number analyzed (Participants) | 282 | 96 | 419 | 206 | 97
  Bowel Problems - 12-months | 7.1 [5.9 to 8.3] | 5.9 [4.4 to 7.4] | 6.2 [5.4 to 7.0] | 9.4 [7.7 to 11.1] | 7.2 [5.6 to 8.8]
  Bowel Problems - 24-months: number analyzed (Participants) | 237 | 80 | 381 | 181 | 82
  Bowel Problems - 24-months | 6.2 [5.3 to 7.1] | 5.0 [3.8 to 6.2] | 5.6 [4.8 to 6.4] | 9.5 [7.5 to 11.5] | 6.1 [4.6 to 7.6]
  Bowel Problems - 36-months: number analyzed (Participants) | 209 | 75 | 330 | 145 | 67
  Bowel Problems - 36-months | 6.9 [5.8 to 8.0] | 5.9 [4.6 to 7.2] | 5.6 [4.7 to 6.5] | 8.4 [6.5 to 10.3] | 5.8 [3.8 to 7.8]
  Bowel Problems - 48-months: number analyzed (Participants) | 190 | 54 | 302 | 141 | 69
  Bowel Problems - 48-months | 7.1 [5.7 to 8.5] | 4.4 [2.7 to 6.1] | 5.3 [4.4 to 6.2] | 7.1 [5.6 to 8.6] | 7.4 [5.2 to 9.6]

2. Primary Outcome: Overall Quality of Life
Description: Short Form-12 (SF12) - Measures health-related quality of life. Consists of Likert response formats that assess overall health, mental health, vitality, social functioning, and whether ones health or pain limits their daily physical activities. The SF-12 also contains four categorical questions (yes or no) that assess limitations in functioning due to physical and emotional health. The SF-12 provides the Mental Component Summary score (MCS) and Physical Component Summary score (PCS), calculated using norm-based scoring, with the mean set at 50 and standard deviation 10. A lower score indicates lower QOL.
Time Frame: 4 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Surveillance | Stereotactic Body Radiation Therapy | Radical Prostatectomy | External Body Radiation Therapy | Brachytherapy
Number analyzed (Participants) | 390 | 104 | 547 | 247 | 125
score on a scale
  Physical Health - Baseline | 47.8 [46.7 to 48.9] | 52.1 [50.5 to 53.7] | 51.1 [50.3 to 51.9] | 47.6 [46.2 to 49.0] | 50.4 [48.8 to 52.0]
  Physical Health - 3-months: number analyzed (Participants) | 306 | 99 | 445 | 224 | 108
  Physical Health - 3-months | 47.6 [46.4 to 48.8] | 50.8 [49.0 to 52.6] | 49.4 [48.5 to 50.3] | 46.4 [45.0 to 47.8] | 49.0 [47.4 to 50.6]
  Physical Health - 12-months: number analyzed (Participants) | 282 | 96 | 419 | 206 | 97
  Physical Health - 12-months | 48.2 [47.1 to 49.3] | 50.8 [49.2 to 52.4] | 49.8 [48.9 to 50.7] | 46.9 [45.5 to 48.3] | 48.7 [46.8 to 50.6]
  Physical Health - 24-months: number analyzed (Participants) | 237 | 80 | 381 | 181 | 82
  Physical Health - 24-months | 46.8 [45.5 to 48.1] | 51.2 [49.3 to 53.1] | 48.6 [47.6 to 49.6] | 46.2 [44.7 to 47.7] | 47.3 [45.1 to 49.5]
  Physical Health - 36-months: number analyzed (Participants) | 209 | 75 | 330 | 145 | 67
  Physical Health - 36-months | 46.8 [45.4 to 48.2] | 50.8 [48.8 to 52.8] | 49.0 [48.0 to 50.0] | 46.6 [44.8 to 48.4] | 48.0 [45.7 to 50.3]
  Physical Health - 48-months: number analyzed (Participants) | 190 | 54 | 302 | 141 | 69
  Physical Health - 48-months | 46.1 [44.7 to 47.5] | 50.7 [48.5 to 52.9] | 48.4 [47.3 to 49.5] | 45.9 [44.2 to 47.6] | 45.8 [43.3 to 48.3]
  Mental Health - Baseline | 54.6 [53.8 to 55.4] | 53.2 [51.7 to 54.7] | 52.0 [51.2 to 52.8] | 52.9 [51.7 to 54.1] | 54.8 [53.3 to 56.3]
  Mental Health - 3-months: number analyzed (Participants) | 306 | 99 | 445 | 224 | 108
  Mental Health - 3-months | 55.0 [54.1 to 55.9] | 54.8 [53.4 to 56.2] | 52.6 [51.7 to 53.5] | 52.9 [51.7 to 54.1] | 53.4 [51.8 to 55.0]
  Mental Health - 12-months: number analyzed (Participants) | 282 | 96 | 419 | 206 | 97
  Mental Health - 12-months | 54.2 [53.2 to 55.2] | 55.2 [53.9 to 56.5] | 54.1 [53.3 to 54.9] | 54.0 [52.8 to 55.2] | 55.6 [54.1 to 57.1]
  Mental Health - 24-months: number analyzed (Participants) | 237 | 80 | 381 | 181 | 82
  Mental Health - 24-months | 55.6 [54.6 to 56.6] | 54.7 [53.1 to 56.3] | 54.1 [53.2 to 55.0] | 54.1 [52.8 to 55.4] | 55.8 [54.2 to 57.4]
  Mental Health - 36-months: number analyzed (Participants) | 209 | 75 | 330 | 145 | 67
  Mental Health - 36-months | 55.3 [54.2 to 56.4] | 54.5 [52.5 to 56.5] | 53.9 [53.0 to 54.8] | 54.2 [52.7 to 55.7] | 55.4 [53.5 to 57.3]
  Mental Health - 48-months: number analyzed (Participants) | 190 | 54 | 302 | 141 | 69
  Mental Health - 48-months | 54.9 [53.8 to 56.0] | 55.1 [53.1 to 57.1] | 54.5 [53.5 to 55.5] | 54.0 [52.5 to 55.5] | 56.2 [54.2 to 58.2]

3. Primary Outcome: Prostate Cancer Recurrence
Description: Percentage of patients who had a recurrence of prostate cancer during 5 years of follow-up.
Time Frame: From date of completion of treatment (radiation or surgery) until the date of recurrence or date of death from any cause, whichever came first, assessed up to 5 years.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiation Therapy | Radical Prostatectomy | External Body Radiation Therapy | Brachytherapy
Number analyzed (Participants) | 104 | 547 | 247 | 125
percentage of participants | 6.7 [3.3 to 13.2] | 13.5 [10.8 to 16.7] | 3.6 [1.7 to 6.8] | 7.2 [2.7 to 13.4]

4. Secondary Outcome: Prostate Cancer Anxiety
Description: Prostate cancer anxiety was measured by the validated Memorial Anxiety Scale for Prostate Cancer (MAX-PC), with 18 questions assessing anxiety related to prostate cancer (11 items, total score 0 to 33), PSA testing (3 items, total score 0 to 9), and fear of recurrence (4 items, total score 0 to 12). The subscale for prostate cancer anxiety asks the patient to report how frequently comments about prostate cancer were true for them during the past week (not at all, rarely, sometimes, or often). The subscale for PSA testing anxiety asks the patient to indicate how frequently situations have ever been true for them. The subscale for anxiety related to prostate cancer recurrence asks the patient to indicate how much they agree or disagree with statements about their own health during the past week. A higher score in each subscale indicates more anxiety.
Time Frame: 4 years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Surveillance | Stereotactic Body Radiation Therapy | Radical Prostatectomy | External Body Radiation Therapy | Brachytherapy
Number analyzed (Participants) | 390 | 104 | 547 | 247 | 125
score on a scale
  Prostate cancer anxiety - 12-months: number analyzed (Participants) | 282 | 96 | 419 | 206 | 97
  Prostate cancer anxiety - 12-months | 1.6 [1.5 to 1.7] | 1.4 [1.3 to 1.5] | 1.6 [1.5 to 1.7] | 1.6 [1.5 to 1.7] | 1.5 [1.4 to 1.6]
  Prostate cancer anxiety - 24-months: number analyzed (Participants) | 237 | 80 | 381 | 181 | 82
  Prostate cancer anxiety - 24-months | 1.5 [1.4 to 1.6] | 1.3 [1.2 to 1.4] | 1.5 [1.4 to 1.6] | 1.5 [1.4 to 1.6] | 1.4 [1.3 to 1.5]
  Prostate cancer anxiety - 36-months: number analyzed (Participants) | 209 | 75 | 330 | 145 | 67
  Prostate cancer anxiety - 36-months | 1.4 [1.3 to 1.5] | 1.3 [1.2 to 1.4] | 1.5 [1.4 to 1.6] | 1.5 [1.4 to 1.6] | 1.3 [1.2 to 1.4]
  Prostate cancer anxiety - 48-months: number analyzed (Participants) | 190 | 54 | 302 | 141 | 69
  Prostate cancer anxiety - 48-months | 1.5 [1.4 to 1.6] | 1.2 [1.1 to 1.6] | 1.5 [1.4 to 1.6] | 1.5 [1.4 to 1.6] | 1.3 [1.2 to 1.4]
  Recurrence anxiety - 12-months: number analyzed (Participants) | 0 | 96 | 419 | 206 | 97
  Recurrence anxiety - 12-months |  | 1.5 [1.4 to 1.6] | 1.7 [1.6 to 1.8] | 1.9 [1.8 to 2.0] | 1.8 [1.7 to 1.9]
  Recurrence anxiety - 24-months: number analyzed (Participants) | 0 | 80 | 381 | 181 | 82
  Recurrence anxiety - 24-months |  | 1.6 [1.5 to 1.7] | 1.7 [1.6 to 1.8] | 1.8 [1.7 to 1.9] | 1.7 [1.6 to 1.8]
  Recurrence anxiety - 36-months: number analyzed (Participants) | 0 | 75 | 330 | 145 | 67
  Recurrence anxiety - 36-months |  | 1.5 [1.4 to 1.6] | 1.7 [1.6 to 1.8] | 1.9 [1.8 to 2.0] | 1.6 [1.5 to 1.7]
  Recurrence anxiety - 48-months: number analyzed (Participants) | 0 | 54 | 302 | 141 | 69
  Recurrence anxiety - 48-months |  | 1.5 [1.4 to 1.6] | 1.7 [1.6 to 1.8] | 1.8 [1.7 to 1.9] | 1.6 [1.5 to 1.7]
  PSA test anxiety - 12-months: number analyzed (Participants) | 282 | 96 | 419 | 206 | 97
  PSA test anxiety - 12-months | 1.2 [1.1 to 1.3] | 1.1 [1.0 to 1.2] | 1.2 [1.2 to 1.2] | 1.2 [1.1 to 1.3] | 1.1 [1.0 to 1.2]
  PSA test anxiety - 24-months: number analyzed (Participants) | 237 | 80 | 381 | 181 | 82
  PSA test anxiety - 24-months | 1.2 [1.1 to 1.3] | 1.1 [1.0 to 1.2] | 1.2 [1.2 to 1.2] | 1.2 [1.1 to 1.3] | 1.1 [1.0 to 1.2]
  PSA test anxiety - 36-months: number analyzed (Participants) | 209 | 75 | 330 | 145 | 67
  PSA test anxiety - 36-months | 1.2 [1.1 to 1.3] | 1.1 [1.0 to 1.2] | 1.2 [1.2 to 1.2] | 1.2 [1.1 to 1.3] | 1.1 [1.0 to 1.2]
  PSA test anxiety - 48-months: number analyzed (Participants) | 190 | 54 | 302 | 141 | 69
  PSA test anxiety - 48-months | 1.2 [1.1 to 1.3] | 1.1 [1.0 to 1.2] | 1.2 [1.2 to 1.2] | 1.2 [1.1 to 1.3] | 1.0 [1.0 to 1.0]

5. Secondary Outcome: Decisional Regret
Description: Decisional regret was measured by a validated scale for prostate cancer. The five items of the decisional regret scale assess (on a Likert scale) a patient's feeling that he chose the wrong treatment, a wish to change the decision, or doubt about treatment value.
  Answers are converted to a score from 0 (no regret) to 100 (maximum regret). Decisional regret provides an assessment of the overall decisional and treatment experience from a patient perspective.
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Surveillance | Stereotactic Body Radiation Therapy | Radical Prostatectomy | External Body Radiation Therapy | Brachytherapy
Number analyzed (Participants) | 390 | 104 | 547 | 247 | 125
percentage of participants
  12-months: number analyzed (Participants) | 261 | 95 | 406 | 193 | 93
  12-months | 9.2 [6.0 to 13.4] | 1.1 [0.0 to 5.7] | 15.0 [11.7 to 18.9] | 8.3 [4.8 to 13.1] | 9.7 [4.5 to 17.6]
  24-months: number analyzed (Participants) | 230 | 79 | 368 | 174 | 77
  24-months | 6.5 [3.7 to 10.5] | 7.6 [2.8 to 15.8] | 18.8 [14.9 to 23.1] | 8.6 [4.9 to 13.8] | 6.5 [2.1 to 14.5]
  36-months: number analyzed (Participants) | 198 | 74 | 316 | 138 | 63
  36-months | 5.6 [2.8 to 9.7] | 9.5 [3.9 to 18.5] | 13.9 [10.3 to 18.2] | 10.1 [5.7 to 16.4] | 9.5 [3.6 to 19.6]
  48-months: number analyzed (Participants) | 186 | 53 | 292 | 136 | 66
  48-months | 5.9 [3.0 to 10.3] | 7.5 [2.1 to 18.2] | 14.0 [10.3 to 18.6] | 12.5 [7.5 to 19.3] | 12.1 [5.4 to 22.5]

6. Secondary Outcome: 5-year Mortality
Description: Percentage of patients who died within 5 years of follow-up.
Time Frame: From date of diagnosis until date of death or end of follow-up up to 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Surveillance | Stereotactic Body Radiation Therapy | Radical Prostatectomy | External Body Radiation Therapy | Brachytherapy
Number analyzed (Participants) | 390 | 104 | 547 | 247 | 125
percentage of participants | 9.5 [6.8 to 12.8] | 2.9 [0.6 to 8.2] | 3.3 [2.0 to 5.2] | 11.3 [7.7 to 16.0] | 4.8 [1.8 to 10.2]

7. Other Pre Specified Outcome: Number of Physician Visits During Follow-up
Description: Number of physician and specialist visits during treatment, subsequent monitoring of recurrence and management of prostate cancer treatment-related morbidity. Assessed through analysis of healthcare claims linked to cohort data.
Time Frame: 4 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: visits
Groups:
- Any Active Treatment: Patients who received initial treatment with surgery or radiation, including brachytherapy or SBRT.
- SBRT/EBRT: Patients who received initial treatment with stereotactic body radiation therapy (SBRT) or external body radiation therapy (EBRT).
Arm/Group | Active Surveillance | Any Active Treatment | Radical Prostatectomy | SBRT/EBRT | Brachytherapy
Number analyzed (Participants) | 88 | 211 | 97 | 79 | 35
visits
  Total prostate cancer visits | 6.1 (3.3) | 4.6 (3.2) | 4.4 (3.4) | 5.0 (3.1) | 4.7 (2.7)
  Total physician visits | 7.6 (3.8) | 6.1 (3.7) | 5.6 (3.9) | 6.8 (3.6) | 6.0 (3.3)
  General practitioner visits | 1.1 (1.4) | 0.8 (1.6) | 0.6 (1.4) | 1.1 (1.7) | 0.9 (1.8)
  Urology/Oncology visits | 5.1 (3.3) | 4.1 (2.6) | 4.0 (2.9) | 4.4 (2.5) | 3.6 (2.2)
  Other specialists visits | 0.1 (0.5) | 0.1 (0.6) | 0.1 (0.7) | 0.1 (0.5) | 0.0 (0.0)

8. Other Pre Specified Outcome: Number of Diagnostic Tests and Procedures During Follow-up
Description: Number of diagnostic tests and procedures including biopsies, radiographic scans, laboratory tests, and procedures to assess cancer progression (active surveillance) or recurrence and work-up for treatment-related morbidity. Assessed through analysis of healthcare claims linked to cohort data.
Time Frame: 4 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: tests or procedures
Arm/Group | Active Surveillance | Any Active Treatment | Radical Prostatectomy | SBRT/EBRT | Brachytherapy
Number analyzed (Participants) | 88 | 211 | 97 | 79 | 35
tests or procedures
  PSA test | 4.6 (2.3) | 4.7 (2.8) | 5.3 (3.2) | 4.3 (2.4) | 4.1 (2.4)
  Other tests and procedures | 1.4 (1.3) | 0.4 (0.6) | 0.2 (0.5) | 0.4 (0.6) | 0.7 (0.7)
  Total tests and procedures | 6.0 (2.7) | 5.1 (2.9) | 5.5 (3.3) | 4.7 (2.4) | 4.8 (2.5)

ADVERSE EVENTS:
Time Frame: 5 years
Description: Serious and other (not including serious) adverse events were not monitored/assessed.
Groups:
- NC ProCESS Cohort: NC ProCESS cohort is a population-based, prospective prostate cancer patient cohort.
Arm/Group | NC ProCESS Cohort
All-Cause Mortality (participants affected / at risk) | 58/1110
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT02564120/Prot_SAP_000.pdf